CLINICAL TRIAL: NCT04761822
Title: Systemic Allergic Reactions to SARS-CoV-2 Vaccination
Brief Title: COVID19 SARS Vaccinations: Systemic Allergic Reactions to SARS-CoV-2 Vaccinations
Acronym: SARS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT COVID-19-004; NIAID CRMS ID#: 38814 (Other: DAIT NIAID)
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: SARS-CoV Infection; COVID-19; Allergic Reaction; Mast Cell Disorder
Keywords: SARS-CoV-2 vaccination; COVID-19 vaccination; Systemic Allergic Reactions to SARS-CoV-2 vaccination
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Hypersensitivity; Mastocytosis | interventions — 2019-nCoV Vaccine mRNA-1273; BNT162 Vaccine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Due to the different dosing schedules for the Pfizer-BioNTech COVID-19 Vaccine and Moderna COVID-19 Vaccine, it will become apparent to both the site staff and study participant which vaccine has been assigned, once their second injection is scheduled. Participants and the staff will be unblinded (unmasked) during the follow-up call 3 days after the second injection when a third appointment (for those who received a placebo injection first) is, or is not (active vaccinations only) scheduled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Moderna COVID-19 Vaccine (Experimental): The Moderna COVID-19 Vaccine (0.5 mL) will be administered intramuscularly in the deltoid, as a series of two doses (0.5 mL each) administered 1 month (28 days) apart.
  Interventions: Biological: Moderna COVID-19 Vaccine
- Pfizer-BioNTech COVID-19 Vaccine (Experimental): The Pfizer-BioNTech COVID-19 Vaccine (0.3 mL) will be administered intramuscularly in the deltoid, as a series of two doses (0.3 mL each) administered 3 weeks (21 days) apart.
  Interventions: Biological: Pfizer-BioNTech COVID-19 Vaccine
- Placebo +Moderna COVID-19 Vaccine (Experimental): Participants will receive placebo as a first dose followed by two doses of their assigned active vaccine at subsequent visits. 0.5 mL of placebo will be administered intramuscularly in the deltoid.
  The placebo dose will be followed by two doses of Moderna COVID-19 Vaccine, with the first dose administered 1 month later. The Moderna COVID-19 Vaccine (0.5 mL) will be administered intramuscularly in the deltoid, as a series of two doses (0.5 mL each) administered 1 month (28 days) apart.
  Interventions: Biological: Moderna COVID-19 Vaccine; Biological: Placebo
- Placebo+Pfizer-BioNTech COVID-19 Vaccine (Experimental): Participants will receive placebo as a first dose followed by two doses of their assigned active vaccine at subsequent visits. 0.3 mL of placebo will be administered intramuscularly in the deltoid.
  The placebo dose will be followed by two doses of Pfizer-BioNTech COVID-19 Vaccine, with the first dose administered 1 month later. The Pfizer-BioNTech COVID-19 Vaccine (0.3 mL) will be administered intramuscularly in the deltoid, as a series of two doses (0.3 mL each) administered 3 weeks (21 days) apart.
  Interventions: Biological: Pfizer-BioNTech COVID-19 Vaccine; Biological: Placebo

INTERVENTIONS:
Biological: Moderna COVID-19 Vaccine — Intramuscular injection
  Other Names: mRNA-1273
  Arms: Moderna COVID-19 Vaccine; Placebo +Moderna COVID-19 Vaccine
Biological: Pfizer-BioNTech COVID-19 Vaccine — Intramuscular injection
  Other Names: BNT162b2
  Arms: Pfizer-BioNTech COVID-19 Vaccine; Placebo+Pfizer-BioNTech COVID-19 Vaccine
Biological: Placebo — Intramuscular injection
  Other Names: sterile, preservative-free 0.9% Sodium Chloride Injection
  Arms: Placebo +Moderna COVID-19 Vaccine; Placebo+Pfizer-BioNTech COVID-19 Vaccine

SUMMARY:
Background: Allergic reactions have been reported to occur after vaccination with both the Pfizer-BioNTech COVID-19 Vaccine and Moderna COVID-19 Vaccine. Allergic reactions range from mild to severe and include life- threatening anaphylactic reactions, although no deaths have been reported with either vaccine.

This study is designed with two principal aims:

* To estimate the proportions of systemic allergic reactions to the Pfizer-BioNTech COVID-19 Vaccine and the Moderna COVID-19 Vaccine in a High-Allergy/Mast Cell Disorder (HA/MCD) population, and
* If the risk in the HA/MCD is demonstrable, to determine whether the proportions are higher in the HA/MCD in comparison to a representative population without severe allergies or mast cell disorders

DETAILED DESCRIPTION:
This is a multicenter, randomized, initially blinded (masked), phase 2 trial to assess SARS-CoV-2 vaccination reactions in two populations:

* One population including individuals with a history of allergic reactions or Mast Cell Disorder (HA/MCD), and
* One comparison population without severe allergies or mast cell disorders.

Approximately 2040 HA/MCD and 1360 comparison participants will be enrolled across participating sites in the United States. Approximately two-thirds of participants enrolled in each of the 2 groups will be female. This is because the vast majority of cases of anaphylaxis to the COVID-19 vaccines have occurred in women. Enrollment of participants who qualify only on the basis of reactions to multiple unrelated drugs will be limited to approximately 300.

Enrollment of the MCD group is anticipated to be at least 200 participants, and not more than 300 participants.

Participants in each population will be randomized 2:2:1:1 to receive the Pfizer-BioNTech COVID-19 Vaccine, Moderna COVID-19 Vaccine, placebo + Pfizer-BioNTech COVID-19 Vaccine, or placebo + Moderna COVID-19 Vaccine, if enrolled in the initial study period under protocol versions 1.0 -4.0. Participants enrolled under protocol version 5.0 will be randomized 2:1 to receive the Pfizer-BioNTech COVID-19 Vaccine or placebo + Pfizer-BioNTech COVID-19 Vaccine. If enrollment under protocol version 5.0 is robust and sustained, the active vaccine randomization may be changed to the Moderna COVID-19 Vaccine.

Participants randomized to one of the placebo groups will receive placebo as a first dose and will receive two doses of their assigned active vaccine at subsequent visits. During the first visit, all participants will be initially-blinded to whether they are receiving placebo or vaccine, and to which vaccine they are receiving (if enrolling under protocol versions 1.0 -4.0).

Due to the different dosing schedules for the Pfizer-BioNTech COVID-19 Vaccine and Moderna COVID-19 Vaccine, it will become apparent to both the site staff and the study participant which vaccine has been assigned, once the second injection visit is scheduled. However, the blind over placebo versus vaccine will remain in effect until after the second visit. During a follow-up call, scheduled 3 days after the second injection, participants will be unblinded as to whether they received placebo or active vaccine.

However under protocol version 5.0, participants will be told if they received placebo as the first injection during the following up conducted 3 days after. Participants in this phase of the study will also know which company's vaccine they are receiving, as the vaccines are anticipated to be used sequentially and will also be noted in the consent form.

Study Duration: Randomized and vaccinated participants will complete study participation in approximately 29 days if vaccinated with the Pfizer-BioNTech COVID-19 Vaccine, 36 days if vaccinated with the Moderna COVID-19 Vaccine. Participants enrolled under protocol versions 1.0 -4.0 will complete study participation in 50 or 64 days if administered placebo before receiving two doses of either the Pfizer-BioNTech COVID-19 Vaccine or the Moderna COVID-19 Vaccine, respectively and participants enrolled under protocol version 5.0 will complete participation in approximately 36 of 43 days, respectively, if they receive placebo first.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for enrollment as study participants:

Both groups (e.g., High-Allergy and Mast Cell Disorder (HA/MCD) Group and Comparison Group):

1. Able to understand and provide informed consent
2. Male or non-pregnant female ≥12 years of age on the date of first study vaccination/placebo administration (protocol versions 1.0 - 4.0) OR male or non-pregnant female 5-17 years of age on the date of first study vaccination/placebo administration (protocol version 5.0)
3. Females of childbearing potential must have a negative pregnancy test prior to the first vaccination and placebo administration, if applicable.

   --If a participant becomes pregnant after receiving a placebo dose but prior to receiving study vaccination, she will be discontinued from the study
4. Females of reproductive potential° and sexually active must agree to use FDA approved methods of birth control for the duration of the study. These include hormonal contraceptives, intrauterine device, double barrier contraception (i.e., condom plus diaphragm), or male partner with documented vasectomy.

   * Menopause is defined as at least 12 consecutive months without menses; if in question, a follicle stimulating hormone of ≥25 U/mL must be documented.
   * Hysterectomy, bilateral oophorectomy, or bilateral tubal ligation must be documented, as applicable; if documented, women with these conditions are not required to use additional contraception.

High-Allergy and Mast Cell Disorder (HA/MCD) Group:

Individuals who meet at least one of the following criteria are eligible for enrollment in the HA/MCD group:

1. History of a severe allergic reaction to food(s), allergen immunotherapy, insect venom(s), or latex with use of epinephrine within the last 15 years
2. History of an Emergency Department visit with convincing evidence of a systemic allergic reaction (consistent with CoFAR Grade 3 or higher) to food(s), allergen immunotherapy, insect venom(s), or latex within the last 15 years
3. History of documented, immediate allergic reactions to 2 or more unrelated drugs within the last 15 years
4. A convincing clinical history, or a history that is accompanied by a positive skin test, of an immediate reaction to a drug, vaccine, or latex within the last 15 years
5. History of physician-diagnosed idiopathic anaphylaxis requiring epinephrine or an Emergency Department visit in the last 15 years
6. History of a physician-diagnosed mast cell disorder (e.g., mastocytosis, mast cell activation syndrome [MCAS], or hereditary alpha-tryptasemia). MCAS must meet consensus criteria as defined below:

   * Criterion A: Typical clinical signs of severe, recurrent (episodic) systemic Mast Cell Activation are present (often in form of anaphylaxis)

     ---Definition of systemic: involving at least 2 organ systems
   * Criterion B: Involvement of Mast Cell (MC) is documented by biochemical studies

     --- Preferred marker: increase in serum tryptase level from the individual's baseline to plus 20% + 2 ng/ml
   * Criterion C: Response of symptoms to therapy with MC-stabilizing agents, drugs directed against MC mediator production or drugs blocking mediator release or effects of MC-derived mediators
   * NOTE: All 3 Mast Cell Activation Syndrome (MCAS) criteria (A + B + C) must be fulfilled to call a condition MCAS.

Comparison Group:

Individuals who meet all of the following criteria are eligible for enrollment in the comparison group:

1. No history of allergic asthma or atopic dermatitis within the last 10 years
2. No history of chronic spontaneous urticaria, or angioedema
3. No history of allergic reactions to foods or insect venoms
4. No history of allergic reactions to drugs or vaccines
5. No history of anaphylaxis
6. No history of a mast cell disorder (e.g., mastocytosis, mast cell activation syndrome [MCAS], or hereditary alpha- tryptasemia)

Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for enrollment as study participants:

1. Inability or unwillingness of a participant and/or parent/legal guardian to give written informed consent and/or assent, as applicable, or to comply with study protocol
2. Weight less than 15 kg (33 lbs)
3. Prior receipt of any doses of the Pfizer-BioNTech coronavirus disease 2019 (COVID-19) Vaccine, Moderna COVID-19 Vaccine, or any other COVID-19 vaccine
4. History of a severe reaction to any component of the Pfizer-BioNTech COVID-19 Vaccine or Moderna COVID-19 Vaccine
5. History of contact dermatitis with confirmed patch test reaction to Prevalence of polyethylene glycol (PEG)
6. History of reaction to Doxil®
7. Known exposure to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and still within the quarantine window
8. Symptoms consistent with acute COVID-19 infection or known COVID-19 infection (positive Polymerase chain reaction [PCR] or antigen test) and still within the quarantine window
9. Have an acute illness, including body temperature greater than 100.4 degrees Fahrenheit, within 14 days of the first study vaccination/placebo administration or 3 days prior to each subsequent vaccination
10. History of autoimmune or other disorders requiring systemic immune modulators
11. History of acute urticaria within 28 days of randomization
12. Pregnant
13. Have received any vaccines within 14 days of the first study vaccination/placebo administration or plan to receive other vaccines during the study period
14. Had any allergen immunotherapy administration within 24 hours prior to vaccination/placebo administration or plan to receive within 24 hours after vaccination/placebo administration
15. Have received a biologic therapy within 6 months of randomization
16. Use of systemic steroids for any reason within 28 days of randomization
17. Use of Zileuton® within 14 days of randomization
18. Use of any monoclonal antibody agent for treatment or prevention of COVID-19 within 3 months of randomization
19. Coronary artery disease, peripheral or cerebral vascular disease, unstable angina, or cardiac arrhythmia, other than supraventricular tachycardia (SVT)
20. Medically unstable hypertension
21. Current use of beta-blockers, angiotensin-converting enzyme (ACE) inhibitors, monoamine oxidase (MAO) inhibitors, tricyclic anti-depressants or other agents that could interfere with the treatment of anaphylaxis, in the opinion of the investigator
22. Unstable asthma within 3 months of randomization or symptomatic asthma on the day of vaccination, as assessed by the site investigator
23. Have past or current medical problems or findings from physical exam or laboratory testing not listed above, which in the opinion of the investigator, may pose additional risks from participation in the study or which may interfere with the ability to comply with study requirements --This includes individuals with underlying conditions or other medications that, in the opinion of the investigator, may increase risk in the event of an anaphylactic reaction or lead to complications following administration of epinephrine

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R. Baker Jr., MD, Study Chair — Mary H. Weiser Food Allergy Center and Michigan Nanotechnology Institute for Medicine and the Biological Sciences; Rebecca S. Gruchalla, MD, PhD, Study Chair — Division of Allergy and Immunology Departments of Internal Medicine and Pediatrics, University of Texas Southwestern; N. Franklin Atkinson Jr., MD, Study Chair — Graduate Training Program in Clinical Investigation Associate TP Director, Allergy-Immunology Johns Hopkins Asthma & Allergy Center
Locations (29):
- United States (29):
  - University of Arizona Health Sciences, College of Medicine Tucson, Department of Medicine, Division of Pulmonary, Allergy, Critical Care and Sleep Medicine, Tucson, Arizona
  - Arkansas Children's, University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California, Los Angeles Medical Center, Los Angeles, California
  - Stanford Medicine, Sean N. Parker Center for Allergy & Asthma Research, Stanford, California
  - National Jewish Health, Denver, Colorado
  - University Health, University of Miami Health System, Miami, Florida
  - University of South Florida Asthma Allergy and Immunology Clinical Research Unit, Tampa, Florida
  - Emory University School of Medicine, Emory Healthcare: Emory Clinic Allergy and Immunology, Atlanta, Georgia
  - Sinus and Allergy Center of Northwestern University, Chicago, Illinois
  - NorthShore University HealthSystem, Dermatology Clinical Trials Unit, Skokie, Illinois
  - University of Iowa Health Care, Iowa City, Iowa
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health, Ann Arbor, Michigan
  - Henry Ford Hospital and Health System, Detroit, Michigan
  - Saint Louis University Care Center for Specialized Medicine, St Louis, Missouri
  - Mount Sinai Hospital, Department of Medicine, Division of Clinical Immunology, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Rochester Regional Health, Rochester, New York
  - North Carolina Translational and Clinical Sciences Institute-Clinical & Translational Research Center (CTRC) at the University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Allergy & Clinical Immunology, Cleveland, Ohio
  - Penn State Health Allergy, Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - University of Virginia Health System: Department of Medicine, Division of Allergy and Immunology, Charlottesville, Virginia
  - Virginia Commonwealth University, Department of Internal Medicine, Division of Rheumatology, Allergy & Immunology, Richmond, Virginia
  - University of Wisconsin Asthma Allergy Pulmonary Research, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Participant level data access and additional relevant materials will be made available upon completion of the trial.
Time Frame: After completion of the trial, within 24 months status post database lock.
Access Criteria: Registration is available for the Immunology Database and Analysis Portal (ImmPort) at: https://www.immport.org/registration. Submit a rationale for the purpose of requesting study data access.
  ImmPort is a long-term archive of clinical and mechanistic data, a National Institute of Allergy and Infectious Diseases Division of Allergy, Immunology and Transplantation (NIAID DAIT)-funded data repository. This archive is in support of the NIH mission to share data with the public. Data shared through ImmPort is provided by NIH-funded programs, other research organizations and individual scientists, ensuring these discoveries will be the foundation of future research.
URL: https://www.immport.org/home

REFERENCES:
- See also: National Institutes of Health News Release Describing Study — https://www.nih.gov/news-events/news-releases/nih-begins-study-allergic-reactions-moderna-pfizer-biontech-covid-19-vaccines
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 746 participants were enrolled across 28 US sites between April 2021 and February 2022. Of those enrolled, 729 participants were randomized and 686 initiated study treatment. The 60 participants who did not initiate study treatment were terminated because they did not meet eligibility criteria, withdrew their consent, or were lost to follow-up.
Pre-assignment Details: Participants were allowed to be randomized up to 14 days prior to their first injection visit to allow for batch scheduling and minimization of vaccine waste. During this time, some participants failed or no longer met eligibility criteria, withdrew their consent, or were lost to follow-up.
Groups:
- Pfizer-BioNTech COVID-19 Vaccine: The Pfizer-BioNTech COVID-19 Vaccine (0.3 mL for those 12 years and older, 0.2 mL for those aged 5 to 11 years) was administered intramuscularly in the deltoid, as a series of two doses (0.3 mL each for those 12 years and older, 0.2 mL for those aged 5 to 11 years), 3 weeks (21 days) apart.
- Moderna COVID-19 Vaccine: The Moderna COVID-19 Vaccine (0.5 mL for those 12 years and older, 0.25 mL for those aged 5 to 11 years) was administered intramuscularly in the deltoid, as a series of two doses (0.5 mL each for those 12 years and older, 0.25 mL each for those aged 5 to 11 years), 1 month (28 days) apart.
- Placebo + Pfizer-BioNTech COVID-19 Vaccine: The placebo dose (0.3 mL for those 12 years and older, 0.2 mL for those aged 5 to 11 years), a sterile, preservative-free 0.9% Sodium Chloride Injection, was administered intramuscularly in the deltoid as a first dose followed by two doses of Pfizer-BioNTech COVID-19 Vaccine starting either 7 or 21 days later, depending upon protocol version. The Pfizer-BioNTech COVID-19 Vaccine (0.3 mL for those 12 years and older, 0.2 mL for those aged 5 to 11 years) was administered intramuscularly in the deltoid, as a series of two doses (0.3 mL each for those 12 years and older, 0.2 mL for those aged 5 to 11 years) administered 3 weeks (21 days) apart.
- Placebo + Moderna COVID-19 Vaccine: The placebo dose (0.5 mL for those 12 years and older, 0.25 mL for those aged 5 to 11 years), a sterile, preservative-free 0.9% Sodium Chloride Injection, was administered intramuscularly in the deltoid as a first dose followed by two doses of Moderna COVID-19 Vaccine starting either 7 or 28 days later, depending upon protocol version. The Moderna COVID-19 Vaccine (0.5 mL for those 12 years and older, 0.25 mL for those aged 5 to 11 years) was administered intramuscularly in the deltoid, as a series of two doses (0.5 mL each for those 12 years and older, 0.25 mL for those aged 5 to 11 years) administered 1 month (28 days) apart.
Period: Overall Study
Arm/Group | Pfizer-BioNTech COVID-19 Vaccine | Moderna COVID-19 Vaccine | Placebo + Pfizer-BioNTech COVID-19 Vaccine | Placebo + Moderna COVID-19 Vaccine
Started | 227 | 219 | 117 | 123
Completed | 219 | 209 | 113 | 105
Not Completed | 8 | 10 | 4 | 18
Not completed — Adverse Event | 3 | 1 | 1 | 3
Not completed — Lost to Follow-up | 1 | 0 | 2 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 8 | 1 | 11
Not completed — Previously rec'd COVID-19 vaccine | 1 | 0 | 0 | 0
Not completed — Participant requested unblinding | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who initiated study treatment.
Groups:
- Placebo + Pfizer-BioNTech COVID-19 Vaccine: The placebo dose (0.3 mL for those 12 years and older, 0.2 mL for those aged 5 to 11 years), a sterile, preservative-free 0.9% Sodium Chloride Injection, was administered intramuscularly in the deltoid as a first dose followed by two doses of Pfizer-BioNTech COVID-19 Vaccine starting either 7 or 21 days later, depending upon protocol version. The Pfizer-BioNTech COVID-19 Vaccine (0.3 mL for those 12 years and older, 0.2 mL for those aged 5 to 11 years) was administered intramuscularly in the deltoid, as a series of two doses (0.3 mL each mL for those 12 years and older, 0.2 mL for those aged 5 to 11 years) administered 3 weeks (21 days) apart.
- Placebo + Moderna COVID-19 Vaccine: The placebo dose (0.5 mL for those 12 years and older, 0.25 mL for those aged 5 to 11 years), a sterile, preservative-free 0.9% Sodium Chloride Injection, was administered intramuscularly in the deltoid as a first dose followed by two doses of Pfizer-BioNTech COVID-19 Vaccine starting either 7 or 28 days later, depending upon protocol version. The Moderna COVID-19 Vaccine (0.5 mL for those 12 years and older, 0.25 mL for those aged 5 to 11 years) was administered intramuscularly in the deltoid, as a series of two doses (0.5 mL each for those 12 years and older, 0.25 mL for those aged 5 to 11 years) administered 1 month (28 days) apart.
- Total: Total of all reporting groups
Arm/Group | Pfizer-BioNTech COVID-19 Vaccine | Moderna COVID-19 Vaccine | Placebo + Pfizer-BioNTech COVID-19 Vaccine | Placebo + Moderna COVID-19 Vaccine | Total
Number analyzed (Participants) | 227 | 219 | 117 | 123 | 686
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33 | 21 | 19 | 18 | 91
  Between 18 and 65 years | 182 | 195 | 95 | 102 | 574
  >=65 years | 12 | 3 | 3 | 3 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (16.97) | 37.7 (15.10) | 35.3 (16.38) | 35.3 (15.89) | 36.9 (16.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 145 | 80 | 80 | 457
  Male | 75 | 74 | 37 | 43 | 229
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 19 | 12 | 15 | 76
  Not Hispanic or Latino | 197 | 199 | 104 | 106 | 606
  Unknown or Not Reported | 0 | 1 | 1 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 0 | 3
  Asian | 18 | 19 | 7 | 8 | 52
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 31 | 33 | 16 | 18 | 98
  White | 151 | 151 | 84 | 87 | 473
  More than one race | 10 | 7 | 3 | 4 | 24
  Unknown or Not Reported | 15 | 9 | 6 | 6 | 36
Region of Enrollment [Number; unit: participants]
  United States | 227 | 219 | 117 | 123 | 686
Cohort [Count of Participants; unit: Participants] — Participants with a history of: severe allergic reaction to food, allergen immunotherapy, insect venom, or latex in the last 15 years; allergic reactions to 2+ unrelated drugs; idiopathic anaphylaxis in the last 15 years; or mast cell disorder comprised the high allergy and mast cell disorder (HA/MCD) cohort. Participants with no history of: allergic asthma or atopic dermatitis in the last 10 years; chronic spontaneous urticaria or angioedema; allergic reaction to food or insect venom, allergic reaction to drugs or vaccines; anaphylaxis; or mast cell disorder comprised the comparison cohort.
  Participants
    HA/MCD | 131 | 118 | 65 | 70 | 384
    Comparison | 96 | 101 | 52 | 53 | 302

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Experienced a Systemic Allergic Reaction (CoFAR Grade 2+ Regardless of Tryptase or CoFAR Grade 1 With Elevated Tryptase) Within 90 Minutes Post-vaccination to Either Dose of Pfizer-BioNTech COVID-19 Vaccine.
Description: Allergic reactions were graded using the Consortium of Food Allergy Research (CoFAR) Grading Scale for Systemic Allergic Reactions, Version 3.0. The scale ranges from grade 1 through 5. The higher the grade, the more severe the allergic reaction. Tryptase is an enzyme released into the blood during an allergic reaction. An elevation in tryptase is defined as a value that is higher than 1.2 x the baseline tryptase plus 2 ng/ml. Subjects who did not receive their second dose of the vaccine were not included unless they reacted (per the endpoint) to the first dose. The comparison is between the High Allergy/Mast Cell Disorder and Comparison populations.
Time Frame: Within the 90-minute post-vaccination observation period to either dose of the Pfizer-BioNTech COVID-19 Vaccine.
Population: Participants who received the Pfizer-BioNTech COVID-19 Vaccine (assigned to Pfizer-BioNTech COVID-19 Vaccine or Placebo + Pfizer-BioNTech COVID-19 Vaccine arms). Participants who did not receive their second dose were not included unless they reacted to the first dose; there were 5 in the HA/MCD group and 4 in the comparison group who were excluded.
Measure: Count of Participants; unit: Participants
Groups:
- Pfizer-BioNTech COVID-19 Vaccine: HA/MCD Cohort: Participants with a history of high allergy/mast cell disorder who received the Pfizer-BioNTech COVID-19 Vaccine (assigned to Pfizer-BioNTech COVID-19 Vaccine or Placebo + Pfizer-BioNTech COVID-19 Vaccine arms). There were 5 participants that did not receive their second dose for reasons other than a reaction to the first dose and were not included.
- Pfizer-BioNTech COVID-19 Vaccine: Comparison Cohort: Participants without a history of high allergy/mast cell disorder who received the Pfizer-BioNTech COVID-19 Vaccine (assigned to Pfizer-BioNTech COVID-19 Vaccine or Placebo + Pfizer-BioNTech COVID-19 Vaccine arms). There were 4 participants that did not receive their second dose for reasons other than a reaction to the first dose and were not included.
Arm/Group | Pfizer-BioNTech COVID-19 Vaccine: HA/MCD Cohort | Pfizer-BioNTech COVID-19 Vaccine: Comparison Cohort
Number analyzed (Participants) | 191 | 144
Participants | 5 | 0
Statistical Analysis 1: Comparison: Pfizer-BioNTech COVID-19 Vaccine: HA/MCD Cohort vs Pfizer-BioNTech COVID-19 Vaccine: Comparison Cohort; The null hypothesis is that the risk difference, where the difference is represented as the high allergy/mast cell disorder cohort proportion minus comparison cohort proportion, is not statistically different from 0 (i.e. there is no difference); Test type: Superiority; p = 0.066, Barnard's Exact Unconditional Test — Two-sided test using the central method of doubling the one-sided p-value; Risk Difference (RD) = 0.026, 95% CI 2-sided [-0.002 to 0.060]

2. Primary Outcome: Proportion of Participants Who Experienced a Systemic Allergic Reaction (CoFAR Grade 2+ Regardless of Tryptase or CoFAR Grade 1 With Elevated Tryptase) Within 90 Minutes Post-vaccination to Either Dose of the Moderna COVID-19 Vaccine.
Description: as for outcome 1
Time Frame: Within the 90-minute post-vaccination observation period to either dose of the Moderna COVID-19 Vaccine.
Population: Participants who received the Moderna COVID-19 Vaccine (assigned to Moderna COVID-19 Vaccine or Placebo + Moderna COVID-19 Vaccine arms). Participants who did not receive their second dose were not included unless they reacted to the first dose; there were 15 in the HA/MCD group and 10 in the comparison group who were excluded.
Measure: Count of Participants; unit: Participants
Groups:
- Moderna COVID-19 Vaccine: HA/MCD Cohort: Participants with a history of high allergy/mast cell disorder who received the Moderna COVID-19 Vaccine (assigned to Moderna COVID-19 Vaccine or Placebo + Moderna COVID-19 Vaccine arms). There were 15 participants that did not receive their second dose for reasons other than a reaction to the first dose and were not included.
- Moderna COVID-19 Vaccine: Comparison Cohort: Participants without a history of high allergy/mast cell disorder who received the Moderna COVID-19 Vaccine (assigned to Moderna COVID-19 Vaccine or Placebo + Moderna COVID-19 Vaccine arms). There were 10 participants that did not receive their second dose for reasons other than a reaction to the first dose and were not included.
Arm/Group | Moderna COVID-19 Vaccine: HA/MCD Cohort | Moderna COVID-19 Vaccine: Comparison Cohort
Number analyzed (Participants) | 173 | 144
Participants | 2 | 0
Statistical Analysis 1: Comparison: Moderna COVID-19 Vaccine: HA/MCD Cohort vs Moderna COVID-19 Vaccine: Comparison Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.267, Barnard's Exact Unconditional Test — Two-sided test using the central method of doubling the one-sided p-value; Risk Difference (RD) = 0.012, 95% CI 2-sided [-0.016 to 0.042]

3. Secondary Outcome: The Proportion of Participants Who Experienced a Severe (CoFAR Grade 3+) Systemic Allergic Reaction Within 90 Minutes Post-vaccination to Either Dose of the Pfizer-BioNTech COVID-19 Vaccine.
Description: Allergic reactions were graded using the Consortium of Food Allergy Research (CoFAR) Grading Scale for Systemic Allergic Reactions, Version 3.0. The scale ranges from grade 1 through 5. The higher the grade, the more severe the allergic reaction. Subjects who did not receive their second dose of the vaccine were not included unless they reacted (per the endpoint) to the first dose. The comparison is between the High Allergy/Mast Cell Disorder and Comparison populations.
Time Frame: Within the 90-minute post-vaccination observation period to either dose of the Pfizer-BioNTech COVID-19 Vaccine.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pfizer-BioNTech COVID-19 Vaccine: HA/MCD Cohort | Pfizer-BioNTech COVID-19 Vaccine: Comparison Cohort
Number analyzed (Participants) | 191 | 144
Participants | 3 | 0
Statistical Analysis 1: Comparison: Pfizer-BioNTech COVID-19 Vaccine: HA/MCD Cohort vs Pfizer-BioNTech COVID-19 Vaccine: Comparison Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.165, Barnard's Exact Unconditional Test — Two-sided test using the central method of doubling the one-sided p-value; Risk Difference (RD) = 0.016, 95% CI 2-sided [-0.011 to 0.046]

4. Secondary Outcome: The Proportion of Participants Who Experienced a Severe (CoFAR Grade 3+) Systemic Allergic Reaction Within the 90-minute Post-vaccination Observation Period to Either Dose of the Moderna COVID-19 Vaccine.
Description: as for outcome 3
Time Frame: Within the 90-minute post-vaccination observation period to either dose of the Moderna COVID-19 Vaccine.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Moderna COVID-19 Vaccine: HA/MCD Cohort | Moderna COVID-19 Vaccine: Comparison Cohort
Number analyzed (Participants) | 173 | 144
Participants | 1 | 0
Statistical Analysis 1: Comparison: Moderna COVID-19 Vaccine: HA/MCD Cohort vs Moderna COVID-19 Vaccine: Comparison Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.572, Barnard's Exact Unconditional Test — Two-sided test using the central method of doubling the one-sided p-value; Risk Difference (RD) = 0.006, 95% CI 2-sided [-0.021 to 0.033]

5. Secondary Outcome: The Proportion of Participants Who Experienced an Anaphylactic Reaction Per Brighton Collaboration Criteria (Levels 1-3) Within 90 Minutes Post-vaccination to Either Dose of the Pfizer-BioNTech COVID-19 Vaccine.
Description: Allergic reactions were graded using the Brighton Collaboration Criteria. The scale ranges from level 1 through 3. Level 1 represents the highest level of diagnostic certainty that a reported case is anaphylaxis, levels 2 and 3 represent successively lower levels of diagnostic certainty. Subjects who did not receive their second dose of the vaccine were not included unless they reacted (per the endpoint) to the first dose. The comparison is between the High Allergy/Mast Cell Disorder and Comparison populations.
Time Frame: Within the 90-minute post-vaccination observation period to either dose of the Pfizer-BioNTech COVID-19 Vaccine.
Population: Participants who received the Pfizer-BioNTech COVID-19 Vaccine (assigned to Pfizer-BioNTech COVID-19 Vaccine or Placebo + Pfizer-BioNTech COVID-19 Vaccine arm). Participants who did not receive their second dose were not included unless they reacted to the first dose; there were 5 in the HA/MCD group and 4 in the comparison group who were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Pfizer-BioNTech COVID-19 Vaccine: HA/MCD Cohort | Pfizer-BioNTech COVID-19 Vaccine: Comparison Cohort
Number analyzed (Participants) | 191 | 144
Participants | 3 | 0
Statistical Analysis 1: Comparison: Pfizer-BioNTech COVID-19 Vaccine: HA/MCD Cohort vs Pfizer-BioNTech COVID-19 Vaccine: Comparison Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.165, Barnard's Exact Unconditional Test; Risk Difference (RD) = 0.016, 95% CI 2-sided [-0.011 to 0.046]

6. Secondary Outcome: The Proportion of Participants Who Experienced an Anaphylactic Reaction Per Brighton Collaboration Criteria (Levels 1-3) Within 90 Minutes Post-vaccination to Either Dose of the Moderna COVID-19 Vaccine.
Description: as for outcome 5
Time Frame: Within the 90-minute post-vaccination observation period to either dose of the Moderna COVID-19 Vaccine.
Population: Participants who received the Moderna COVID-19 Vaccine (assigned to Moderna COVID-19 Vaccine or Placebo + Moderna COVID-19 Vaccine arm). Participants who did not receive their second dose were not included unless they reacted to the first dose; there were 15 in the HA/MCD group and 10 in the comparison group who were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Moderna COVID-19 Vaccine: HA/MCD Cohort | Moderna COVID-19 Vaccine: Comparison Cohort
Number analyzed (Participants) | 173 | 144
Participants | 1 | 0
Statistical Analysis 1: Comparison: Moderna COVID-19 Vaccine: HA/MCD Cohort vs Moderna COVID-19 Vaccine: Comparison Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.572, Barnard's Exact Unconditional Test — Two-sided test using the central method of doubling the one-sided p-value; Risk Difference (RD) = 0.006, 95% CI 2-sided [-0.021 to 0.033]

7. Secondary Outcome: Proportion of Participants Who Experienced a Systemic Allergic Reaction (CoFAR Grade 2+ Regardless of Tryptase or CoFAR Grade 1 With Elevated Tryptase) Within 90 Minutes Post-vaccination to the First Dose of the Pfizer-BioNTech COVID-19 Vaccine.
Description: Allergic reactions were graded using the Consortium of Food Allergy Research (CoFAR) Grading Scale for Systemic Allergic Reactions, Version 3.0. The scale ranges from grade 1 through 5. The higher the grade, the more severe the allergic reaction. Tryptase is an enzyme released into the blood during an allergic reaction. An elevation in tryptase is defined as a value that is higher than 1.2 x the baseline tryptase plus 2 ng/ml. The comparison is between the participants who received active vaccine as their first, fully blinded, injection (assigned to the Pfizer-BioNTech COVID-19 Vaccine arm) and participants who received their first active vaccine as their second injection (assigned to the Placebo + Pfizer-BioNTech COVID-19 Vaccine arm). Due to the design of the trial, participants would have understood that the second dose in any arm must be an active vaccination.
Time Frame: Within the 90-minute post-vaccination observation period to the first dose of the Pfizer-BioNTech COVID-19 Vaccine.
Population: Participants who received the Pfizer-BioNTech COVID-19 Vaccine (assigned to Pfizer-BioNTech COVID-19 Vaccine or Placebo + Pfizer-BioNTech COVID-19 Vaccine arm). Participants were only included from the HA/MCD cohort. One participant in the Placebo + Pfizer-BioNTech COVID-19 Vaccine arm was not included as they did not receive any active doses.
Measure: Count of Participants; unit: Participants
Groups:
- Pfizer-BioNTech COVID-19 Vaccine First Active Dose: HA/MCD Cohort: Participants with a history of high allergy/mast cell disorder who received the first active dose of Pfizer-BioNTech COVID-19 Vaccine as their first injection (assigned to Pfizer-BioNTech COVID-19 Vaccine).
- Placebo + Pfizer-BioNTech COVID-19 Vaccine First Active Dose: HA/MCD Cohort: Participants with a history of high allergy/mast cell disorder who received the first active dose of Pfizer-BioNTech COVID-19 Vaccine as their second injection (assigned to Placebo + Pfizer-BioNTech COVID-19 Vaccine arm). One participant was not included as they did not receive any active doses.
Arm/Group | Pfizer-BioNTech COVID-19 Vaccine First Active Dose: HA/MCD Cohort | Placebo + Pfizer-BioNTech COVID-19 Vaccine First Active Dose: HA/MCD Cohort
Number analyzed (Participants) | 131 | 64
Participants | 2 | 0
Statistical Analysis 1: Comparison: Pfizer-BioNTech COVID-19 Vaccine First Active Dose: HA/MCD Cohort vs Placebo + Pfizer-BioNTech COVID-19 Vaccine First Active Dose: HA/MCD Cohort; The null hypothesis is that the risk difference, where the difference is represented as the participants that received their first active dose as their first injection proportion minus the participants that received their first active dose as their second injection proportion, is not statistically different from 0 (i.e. there is no difference); Test type: Superiority; p = 0.4574, Barnard's Exact Unconditional Test — Two-sided test using the central method of doubling the one-sided p-value; Risk Difference (RD) = 0.015, 95% CI 2-sided [-0.045 to 0.055]

8. Secondary Outcome: Proportion of Participants Who Experienced a Systemic Allergic Reaction (CoFAR Grade 2+ Regardless of Tryptase or CoFAR Grade 1 With Elevated Tryptase) Within 90 Minutes Post-vaccination to the First Dose of the Moderna COVID-19 Vaccine.
Description: Allergic reactions were graded using the Consortium of Food Allergy Research (CoFAR) Grading Scale for Systemic Allergic Reactions, Version 3.0. The scale ranges from grade 1 through 5. The higher the grade, the more severe the allergic reaction. Tryptase is an enzyme released into the blood during an allergic reaction. An elevation in tryptase is defined as a value that is higher than 1.2 x the baseline tryptase plus 2 ng/ml. The comparison is between the participants who received active vaccine as their first, fully blinded, injection (assigned to the Moderna COVID-19 Vaccine arm) and participants who received their first active vaccine as their second injection (assigned to the Placebo + Moderna COVID-19 Vaccine arm). Due to the design of the trial, participants would have understood that the second dose in any arm must be an active vaccination.
Time Frame: Within the 90-minute post-vaccination observation period to the first dose of the Moderna COVID-19 Vaccine.
Population: Participants who received the Moderna COVID-19 Vaccine (assigned to Moderna COVID-19 Vaccine or Placebo + Moderna COVID-19 Vaccine arms). Participants were only included from the HA/MCD cohort. Six participants in the Placebo + Moderna COVID-19 Vaccine arm were not included as they did not receive any active doses.
Measure: Count of Participants; unit: Participants
Groups:
- Moderna COVID-19 Vaccine First Active Dose: HA/MCD Cohort: Participants with a history of high allergy/mast cell disorder who received the first active dose of Moderna COVID-19 Vaccine as their first injection (assigned to Moderna COVID-19 Vaccine arm).
- Placebo + Moderna COVID-19 Vaccine First Active Dose: HA/MCD Cohort: Participants with a history of high allergy/mast cell disorder who received the first active dose of Moderna COVID-19 Vaccine as their second injection (assigned to Placebo + Moderna COVID-19 Vaccine arm). Six participants were not included as they did not receive any active doses.
Arm/Group | Moderna COVID-19 Vaccine First Active Dose: HA/MCD Cohort | Placebo + Moderna COVID-19 Vaccine First Active Dose: HA/MCD Cohort
Number analyzed (Participants) | 118 | 64
Participants | 0 | 1
Statistical Analysis 1: Comparison: Moderna COVID-19 Vaccine First Active Dose: HA/MCD Cohort vs Placebo + Moderna COVID-19 Vaccine First Active Dose: HA/MCD Cohort; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.3242, Barnard's Exact Unconditional Test — Two-sided test using the central method of doubling the one-sided p-value; Risk Difference (RD) = -0.016, 95% CI 2-sided [-0.086 to 0.018]

9. Secondary Outcome: Proportion of Participants Who Experienced a Systemic Allergic Reaction (CoFAR Grade 2+ Regardless of Tryptase or CoFAR Grade 1 With Elevated Tryptase) Within 90 Minutes Post-vaccination to the Second Dose of the Pfizer-BioNTech COVID-19 Vaccine.
Description: Allergic reactions were graded using the Consortium of Food Allergy Research (CoFAR) Grading Scale for Systemic Allergic Reactions, Version 3.0. The scale ranges from grade 1 through 5. The higher the grade, the more severe the allergic reaction. Tryptase is an enzyme released into the blood during an allergic reaction. An elevation in tryptase is defined as a value that is higher than 1.2 x the baseline tryptase plus 2 ng/ml. The comparison is between the participants who received the second active vaccine as their second injection (assigned to the Pfizer-BioNTech COVID-19 Vaccine arm) and participants who received the second active vaccine as their third injection (assigned to the Placebo + Pfizer-BioNTech COVID-19 Vaccine arm). This comparison is conditional on there being no systemic allergic reaction to the first dose.
Time Frame: Within the 90-minute post-vaccination observation period to the second dose of the Pfizer-BioNTech COVID-19 Vaccine.
Population: Participants from the HA/MCD cohort who received the Pfizer-BioNTech COVID-19 Vaccine (assigned to Pfizer-BioNTech COVID-19 Vaccine or Placebo + Pfizer-BioNTech COVID-19 Vaccine arm). Five (2 reaction to first dose, 3 missing second dose) and 1 (1 reaction to placebo dose) were excluded, respectively.
Measure: Count of Participants; unit: Participants
Groups:
- Pfizer-BioNTech COVID-19 Vaccine Second Active Dose: HA/MCD Cohort: Participants with a history of high allergy/mast cell disorder who received the second active dose of Pfizer-BioNTech COVID-19 Vaccine as their second injection (assigned to Pfizer-BioNTech COVID-19 Vaccine arm). Five participants were not included (2 reacted to first dose, 3 missing second dose).
- Placebo + Pfizer-BioNTech COVID-19 Vaccine Second Active Dose: HA/MCD Cohort: Participants with a history of high allergy/mast cell disorder who received the second active dose of Pfizer-BioNTech COVID-19 Vaccine as their third injection (assigned to Placebo + Pfizer-BioNTech COVID-19 Vaccine arm). One participant was not included as they did not receive any active doses.
Arm/Group | Pfizer-BioNTech COVID-19 Vaccine Second Active Dose: HA/MCD Cohort | Placebo + Pfizer-BioNTech COVID-19 Vaccine Second Active Dose: HA/MCD Cohort
Number analyzed (Participants) | 126 | 64
Participants | 3 | 0
Statistical Analysis 1: Comparison: Pfizer-BioNTech COVID-19 Vaccine Second Active Dose: HA/MCD Cohort vs Placebo + Pfizer-BioNTech COVID-19 Vaccine Second Active Dose: HA/MCD Cohort; The null hypothesis is that the risk difference, where the difference is represented as the participants that received their second active dose as their second injection proportion minus the participants that received their second active dose as their third injection proportion, is not statistically different from 0 (i.e. there is no difference); Test type: Superiority; p = 0.3100, Barnard's Exact Unconditional Test — Two-sided test using the central method of doubling the one-sided p-value; Risk Difference (RD) = 0.024, 95% CI 2-sided [-0.037 to 0.070]

10. Secondary Outcome: Proportion of Participants Who Experienced a Systemic Allergic Reaction (CoFAR Grade 2+ Regardless of Tryptase or CoFAR Grade 1 With Elevated Tryptase) Within 90 Minutes Post-vaccination to the Second Dose of the Moderna COVID-19 Vaccine.
Description: Allergic reactions were graded using the Consortium of Food Allergy Research (CoFAR) Grading Scale for Systemic Allergic Reactions, Version 3.0. The scale is ranges from grade 1 through 5. The higher the grade, the more severe the allergic reaction. Tryptase is an enzyme released into the blood during an allergic reaction. An elevation in tryptase is defined as a value that is higher than 1.2 x the baseline tryptase plus 2 ng/ml. The comparison is between the participants who received the second active vaccine as their second injection (assigned to the Moderna COVID-19 Vaccine arm) and participants who received the second active vaccine as their third injection (assigned to the Placebo + Moderna COVID-19 Vaccine arm). This comparison is conditional on there being no systemic allergic reaction to the first dose.
Time Frame: Within the 90-minute post-vaccination observation period to the second dose of the Moderna COVID-19 Vaccine.
Population: Participants from the HA/MCD cohort who received the Moderna COVID-19 Vaccine (assigned to Moderna COVID-19 Vaccine or Placebo + Moderna COVID-19 Vaccine arm). Six (all missing second dose) and 6 (all missing second dose) were excluded, respectively.
Measure: Count of Participants; unit: Participants
Groups:
- Moderna COVID-19 Vaccine Second Active Dose: HA/MCD Cohort: Participants with a history of high allergy/mast cell disorder who received the second active dose of Moderna COVID-19 Vaccine as their second injection (assigned Moderna COVID-19 Vaccine arm). Six participants were not included due to missing second dose.
- Placebo + Moderna COVID-19 Vaccine Second Active Dose: HA/MCD Cohort: Participants with a history of high allergy/mast cell disorder who received the second active dose of Moderna COVID-19 Vaccine as their third injection (assigned to Placebo + Moderna COVID-19 Vaccine arm). Six participants were not included as they did not receive second doses.
Arm/Group | Moderna COVID-19 Vaccine Second Active Dose: HA/MCD Cohort | Placebo + Moderna COVID-19 Vaccine Second Active Dose: HA/MCD Cohort
Number analyzed (Participants) | 112 | 64
Participants | 1 | 1
Statistical Analysis 1: Comparison: Moderna COVID-19 Vaccine Second Active Dose: HA/MCD Cohort vs Placebo + Moderna COVID-19 Vaccine Second Active Dose: HA/MCD Cohort; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.8070, Barnard's Exact Unconditional Test — Two-sided test using the central method of doubling the one-sided p-value; Risk Difference (RD) = -0.007, 95% CI 2-sided [-0.0783 to 0.0366]

11. Secondary Outcome: The Proportion of Participants Who Experienced a Systemic Allergic Reaction (CoFAR Grade 2+ Regardless of Tryptase or CoFAR Grade 1 With Elevated Tryptase) Within 90 Minutes Post-vaccination to the First Dose, Adjusting for Placebo.
Description: Allergic reactions were graded using the Consortium of Food Allergy Research (CoFAR) Grading Scale for Systemic Allergic Reactions, Version 3.0. The scale ranges from grade 1 through 5. The higher the grade, the more severe the allergic reaction. Tryptase is an enzyme released into the blood during an allergic reaction. An elevation in tryptase is defined as a value that is higher than 1.2 x the baseline tryptase plus 2 ng/ml. The comparison is between participants who had placebo as their first injection (either vaccine) and participants who had Pfizer-BioNTech COVID-19 Vaccine as their first injection. The comparison only includes subjects in the HA/MCD cohort.
Time Frame: Within the 90-minute post-vaccination observation period to the first injection (placebo or active).
Population: Participants who received placebo as their first injection (assigned to Placebo + Pfizer-BioNTech COVID-19 Vaccine arm or Placebo + Moderna COVID-19 Vaccine arm) or received Pfizer-BioNTech COVID-19 Vaccine as their first dose (Pfizer-BioNTech COVID-19 Vaccine arm). Participants were only included from the HA/MCD cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo First Injection: HA/MCD: Participants with a history of high allergy/mast cell disorder who received placebo as their first injection (assigned to Placebo + Pfizer-BioNTech COVID-19 Vaccine arm or Placebo + Moderna COVID-19 Vaccine arm)
- Pfizer-BioNTech COVID-19 Vaccine First Injection: HA/MCD: Participants with a history of high allergy/mast cell disorder who received the active injection of Pfizer-BioNTech COVID-19 Vaccine as their first injection (assigned to Pfizer-BioNTech COVID-19 Vaccine).
Arm/Group | Placebo First Injection: HA/MCD | Pfizer-BioNTech COVID-19 Vaccine First Injection: HA/MCD
Number analyzed (Participants) | 135 | 131
Participants | 2 | 2
Statistical Analysis 1: Comparison: Placebo First Injection: HA/MCD vs Pfizer-BioNTech COVID-19 Vaccine First Injection: HA/MCD; The null hypothesis is that the risk difference, where the difference is represented as the Pfizer-BioNTech COVID-19 vaccine first injection proportion minus comparison placebo first injection proportion, is not statistically different from 0 (i.e. there is no difference); Test type: Superiority; p = 1.000, Barnard's Exact Unconditional Test — Two-sided test using the central method of doubling the one-sided p-value; Risk Difference (RD) = 0.001, 95% CI 2-sided [-0.040 to 0.042]

12. Secondary Outcome: The Proportion of Participants Who Experienced a Systemic Allergic Reaction (CoFAR Grade 2+ Regardless of Tryptase or CoFAR Grade 1 With Elevated Tryptase) Within 90 Minutes Post-vaccination to the First Dose, Adjusting for Placebo.
Description: Allergic reactions were graded using the Consortium of Food Allergy Research (CoFAR) Grading Scale for Systemic Allergic Reactions, Version 3.0. The scale is ranges from grade 1 through 5. The higher the grade, the more severe the allergic reaction. Tryptase is an enzyme released into the blood during an allergic reaction. An elevation in tryptase is defined as a value that is higher than 1.2 x the baseline tryptase plus 2 ng/ml. The comparison is between participants who had placebo as their first injection and participants who had Moderna COVID-19 Vaccine as their first injection. The comparison only includes subjects in the HA/MCD cohort.
Time Frame: Within the 90-minute post-vaccination observation period to the first injection.
Population: Participants who received placebo as their first injection (assigned to Placebo + Pfizer-BioNTech COVID-19 Vaccine arm or Placebo + Moderna COVID-19 Vaccine arm) or received Moderna COVID-19 Vaccine as their first injection (Moderna COVID-19 Vaccine arm). Participants were only included from the HA/MCD cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Moderna COVID-19 Vaccine First Injection: HA/MCD: Participants with a history of high allergy/mast cell disorder who received the active dose of Moderna COVID-19 Vaccine as their first injection (assigned to Moderna COVID-19 Vaccine).
Arm/Group | Placebo First Injection: HA/MCD | Moderna COVID-19 Vaccine First Injection: HA/MCD
Number analyzed (Participants) | 135 | 118
Participants | 2 | 0
Statistical Analysis 1: Comparison: Placebo First Injection: HA/MCD vs Moderna COVID-19 Vaccine First Injection: HA/MCD; The null hypothesis is that the risk difference, where the difference is represented as the Moderna COVID-19 vaccine first injection proportion minus comparison placebo first injection proportion, is not statistically different from 0 (i.e. there is no difference); Test type: Superiority; p = 0.250, Barnard's Exact Unconditional Test — Two-sided test using the central method of doubling the one-sided p-value; Risk Difference (RD) = -0.015, 95% CI 2-sided [-0.053 to 0.018]

13. Secondary Outcome: The Proportion of Participants Who Experienced a Systemic Allergic Reaction (CoFAR Grade 2+) Within 48-hours Post-vaccination to Either Dose of the Pfizer-BioNTech COVID-19 Vaccine.
Description: as for outcome 3
Time Frame: After the 90 minute observation period to 48-hours post-vaccination to either dose of the Pfizer-BioNTech COVID-19 Vaccine.
Population: Participants who received the Pfizer-BioNTech COVID-19 Vaccine (assigned to Pfizer-BioNTech COVID-19 Vaccine or Placebo + Pfizer-BioNTech COVID-19 Vaccine arm). Participants who did not receive their second dose were not included unless they reacted to the first dose; there were 6 in the HA/MCD group and 4 in the comparison group who were excluded.
Measure: Count of Participants; unit: Participants
Groups:
- Pfizer-BioNTech COVID-19 Vaccine: HA/MCD Cohort: Participants with a history of high allergy/mast cell disorder who received the Pfizer-BioNTech COVID-19 Vaccine (assigned to Pfizer-BioNTech COVID-19 Vaccine or Placebo + Pfizer-BioNTech COVID-19 Vaccine arms). There were 6 participants that did not receive their second dose for reasons other than a reaction to the first dose and were not included.
Arm/Group | Pfizer-BioNTech COVID-19 Vaccine: HA/MCD Cohort | Pfizer-BioNTech COVID-19 Vaccine: Comparison Cohort
Number analyzed (Participants) | 190 | 144
Participants | 11 | 0
Statistical Analysis 1: Comparison: Pfizer-BioNTech COVID-19 Vaccine: HA/MCD Cohort vs Pfizer-BioNTech COVID-19 Vaccine: Comparison Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.004, Barnard's Exact Unconditional Test — Two-sided test using the central method of doubling the one-sided p-value; Risk Difference (RD) = 0.058, 95% CI 2-sided [0.024 to 0.101]

14. Secondary Outcome: The Proportion of Participants Who Experienced a Systemic Allergic Reaction (CoFAR Grade 2+) Within 48-hours Post-vaccination to Either Dose of the Moderna COVID-19 Vaccine.
Description: as for outcome 3
Time Frame: After the 90 minute observation period to 48-hours post-vaccination to either dose of the Moderna COVID-19 Vaccine.
Population: Participants who received the Moderna COVID-19 Vaccine (assigned to Moderna COVID-19 Vaccine or Placebo + Moderna COVID-19 Vaccine arm). Participants who did not receive their second dose were not included unless they reacted to the first dose; there were 14 in the HA/MCD group and 10 in the comparison group who were excluded.
Measure: Count of Participants; unit: Participants
Groups:
- Moderna COVID-19 Vaccine: HA/MCD Cohort: Participants with a history of high allergy/mast cell disorder who received the Moderna COVID-19 Vaccine (assigned to Moderna COVID-19 Vaccine or Placebo + Moderna COVID-19 Vaccine arms). There were 14 participants that did not receive their second dose for reasons other than a reaction to the first dose and were not included.
Arm/Group | Moderna COVID-19 Vaccine: HA/MCD Cohort | Moderna COVID-19 Vaccine: Comparison Cohort
Number analyzed (Participants) | 174 | 144
Participants | 13 | 0
Statistical Analysis 1: Comparison: Moderna COVID-19 Vaccine: HA/MCD Cohort vs Moderna COVID-19 Vaccine: Comparison Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Barnard's Exact Unconditional Test — Two-sided test using the central method of doubling the one-sided p-value; Risk Difference (RD) = 0.075, 95% CI 2-sided [0.039 to 0.124]

ADVERSE EVENTS:
Time Frame: From start of study through end of study (up to 64 days).
Arm/Group | Pfizer-BioNTech COVID-19 Vaccine | Moderna COVID-19 Vaccine | Placebo + Pfizer-BioNTech COVID-19 Vaccine | Placebo + Moderna COVID-19 Vaccine
All-Cause Mortality (participants affected / at risk) | 0/227 | 0/219 | 0/117 | 0/123
Serious Adverse Events (participants affected / at risk) | 5/227 | 2/219 | 2/117 | 3/123
Other Adverse Events (participants affected / at risk) | 185/227 | 195/219 | 100/117 | 104/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pfizer-BioNTech COVID-19 Vaccine (N=227) | Moderna COVID-19 Vaccine (N=219) | Placebo + Pfizer-BioNTech COVID-19 Vaccine (N=117) | Placebo + Moderna COVID-19 Vaccine (N=123)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Amoebiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pfizer-BioNTech COVID-19 Vaccine (N=227) | Moderna COVID-19 Vaccine (N=219) | Placebo + Pfizer-BioNTech COVID-19 Vaccine (N=117) | Placebo + Moderna COVID-19 Vaccine (N=123)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mast cell activation syndrome (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Swelling of eyelid (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Visual field defect (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lip erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Oesophageal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (2) | 1 (1) | 3 (3) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Facial discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 4 (5) | 5 (7) | 3 (4)
Feeling abnormal (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Sensation of foreign body (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination site reaction (General disorders) | 131 (242) | 143 (255) | 74 (133) | 69 (130)
Vessel puncture site bruise (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 25 (44) | 25 (31) | 15 (35) | 16 (31)
Milk allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 153 (357) | 163 (378) | 83 (276) | 89 (260)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophil count abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Eosinophil count increased (Investigations) | 4 (4) | 2 (2) | 2 (2) | 2 (4)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemoglobin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 14 (15) | 17 (20) | 9 (11) | 3 (4)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 8 (8) | 7 (7) | 3 (4) | 4 (4)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Mean cell haemoglobin concentration decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Monocyte count increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neutrophil count abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 6 (7) | 4 (6) | 3 (5)
Platelet count decreased (Investigations) | 1 (1) | 2 (3) | 1 (2) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 4 (4) | 4 (6) | 5 (5) | 3 (4)
White blood cell count increased (Investigations) | 3 (3) | 6 (6) | 3 (3) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (7) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 6 (7) | 3 (3) | 4 (6) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurological symptom (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 3 (3) | 2 (2) | 2 (3) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cystitis interstitial (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premenstrual pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (3) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 4 (5) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 11 (17) | 8 (13) | 5 (9) | 5 (12)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (3) | 1 (1)
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Knee operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 6 (7) | 2 (3) | 2 (2) | 5 (6)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT04761822/Prot_003.pdf
  • Statistical Analysis Plan (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT04761822/SAP_001.pdf
  • Informed Consent Form (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT04761822/ICF_002.pdf